CLINICAL TRIAL: NCT02822924
Title: Prostate Artery Embolization for Symptomatic Benign Prostatic Hyperplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Simon Yu, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VIR-13-05
Record Dates: First submitted 2016-06-28; First posted 2016-07-06 (Estimated); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Benign Prostate Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prostate artery embolization treatment (Other): Prostatic artery embolization (PAE) as a new treatment technology is a potentially promising, minimally invasive alternative procedure for BPH, which has been shown to be safe and effective in both animal models and clinical trials.
  Interventions: Procedure: Prostate artery embolization (PAE)

INTERVENTIONS:
Procedure: Prostate artery embolization (PAE) — Right femoral arterial puncture is performed under local anesthesia. The blood supply to the prostate is mapped by angiography of the iliac vessels and the prostate arteries. Microcatheters are used for super-selective catheterization of the right and left inferior vesicle arteries. Embolization is performed with a microcatheter to deliver microspheres of 300 micron diameter. The microsphere mixture is slowly injected under fluoroscopic guidance. The endpoint of embolization is flow stasis in the prostatic vessels with prostatic gland opacification, without reflux of the mixture to undesired arteries.

SUMMARY:
The objective is to evaluate the clinical effectiveness and safety of PAE in treating patients with BPH.

DETAILED DESCRIPTION:
Benign prostatic hyperplasia (BPH), non-malignant enlargement of the prostate, is a common condition among elderly men with a prevalence increasing with age. When sufficiently large, the hyperplastic nodules compress the urethral canal to cause obstruction of the urethra and interfere the normal flow of urine, leading to symptoms of urinary hesitancy, frequent urination, increased risk of urinary tract infections and urinary retention. While medication is often prescribed as the first treatment option, it often does not adequately restore normal urine flow. Many patients being treated with medication may not achieve sustained improvement in symptoms, or they may stop taking the medication because of side effects, therefore other forms of treatments may be necessary. Although surgery with transurethral resection of prostate (TURP) is a benchmark for BPH treatment, it involves insertion of an endoscope is inserted through the penis, and removal of the prostate piece by piece. While considered a safe technique with a mortality rate below 0.25%, it is not without adverse events. The most frequent complications are ejaculatory disorders (up to 80%), early urinary incontinence (30 to 40%), acute urinary retention caused by blood clots (2 to 5%), sexual impotence (up to 5%), and the need for blood transfusions (0.4 to 7%). Patients who have undergone TURP require surgical retreatment for lower urinary tract symptoms in 3 to 14.5% of cases. Others include infection and urethral stricture. Therefore TURP is only recommended for complicated or severe BPH due to its adverse effects. Prostatic artery embolization (PAE) is a potentially promising, minimally invasive alternative procedure for BPH. Results from early studies showed that PAE might be a safe and effective treatment for BPH.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 50 and 80 years old.
2. Suffered from lower urinary tract symptoms with International Prostate Symptom Score (IPSS) ≥13, despite medical treatment with alpha-blockers for at least 6 months, or
3. Suffered from lower urinary tract symptoms with International Prostate Symptom Score (IPSS) ≥13, for whom medication is contraindicated, not tolerated or refused, or
4. Patients with history of acute retention of urine with or without previous treatment with Alpha-blockers.
5. Patients with QOL score ≥3.
6. Patients with Urine flow rate < 15ml/second or acute urinary retention.
7. Patients with evidence of prostatic enlargement determined by digital rectal examination or ultrasonography (USG), with a prostate size of not less than 40 grams.

Exclusion Criteria:

1. Active urinary tract infection
2. Biopsy proven prostate or bladder cancer, or any recent cancer within 5 years other than basal or squamous cell skin cancer
3. Bladder atonia, neurogenic bladder disorder or other neurological disorder that is impacting bladder function (e.g. multiple sclerosis, Parkinson's disease, spinal cord injuries, etc)
4. Urethral stricture, bladder neck contracture, sphincter abnormalities, urinary obstruction due to causes other than BPH, or other potentially confounding bladder or urethral disease or condition
5. Prostate size <40 grams on CT or MRI
6. Previous non-medical BPH treatment, including surgery, TURP, needle ablation, microwave or laser therapy, balloon dilation, stent implantation, or any other invasive treatment to the prostate
7. Any known condition that limits catheter-based intervention or is a contraindication to embolization, such as intolerance to a vessel occlusion procedure or severe atherosclerosis.
8. Unable to have MRI imaging (e.g. metal implant including pacemaker, replacement joint, etc)
9. Cardiac condition including congestive heart failure or arrhythmia, uncontrolled diabetes mellitus, significant respiratory disease or known immunosuppression which required hospitalization within the previous 6 months
10. Baseline serum creatinine level > 160 umol/L
11. Known upper tract renal disease
12. Cystolithiasis or chronic hematuria within 3 months prior to study treatment
13. Active prostatitis
14. Previous rectal surgery other than hemorrhoidectomy, or history of rectal disease
15. History of pelvic irradiation or radical pelvic surgery
16. Coagulation disturbances not normalized by medical treatment
17. Known major iliac arterial occlusive disease
18. Allergy to iodinated contrast agents
19. Hypersensitivity to gelatin products

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2013-10-07 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
successful procedure | within 1 hour after PAE procedure
  Procedure success defined as technically successful selective prostatic arterial catheterization and embolization

SECONDARY OUTCOMES:
Incidence of procedure related complication | 6-8 hours after treatment until 1 month time
  Complication after treatment procedure will be recorded. Major adverse events, which included ischemic, infectious, or puncture site complications, pain will be recorded and evaluated. Further imaging or laboratory studies are conducted when a complication was suspected.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Yu, Profesor, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Imaging and Interventional Radiology, Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No